CLINICAL TRIAL: NCT06439056
Title: An Open, Single Ascending Dose, Phase 1 Study to Assess the Pharmacokinetics, Safety, and Tolerability of NEX-22A, a Subcutaneous Prolonged-release Injection, in Male and Female Participants With Type 2 Diabetes
Brief Title: Phase 1 Study Assessing the Pharmacokinetics of NEX-22A in Subjects With T2D
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nanexa AB (Industry)
Collaborators: Profil Institut für Stoffwechselforschung GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEX-22-01
Record Dates: First submitted 2024-05-16; First posted 2024-06-03 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; PK study; Long acting injectable; Liraglutid; GLP-1
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Single ascending dose study including 3 cohorts (3 patients/cohort). The subjects will be enrolled in the respective cohorts, starting with cohort 1. NEX-22A will be administered in a sentinel fashion within the cohorts. A single participant will be dosed first in every cohort. If there are no safety concerns as judged by the investigator, the remaining subjects will be dosed at least 10 days after the sentinel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single dose of NEX-22-01 (Experimental): The trial is single ascending dose study where the dose is escalated depending on previous cohorts PK data.
  Interventions: Drug: NEX-22A, a prolonged release formulation of liraglutide

INTERVENTIONS:
Drug: NEX-22A, a prolonged release formulation of liraglutide — NEX-22A, a prolonged release formulation of liraglutide

SUMMARY:
The purpose with the study is to assess pharmacokinetics of NEX-22A in patients with type 2 diabetes.

DETAILED DESCRIPTION:
The trial is a single-centre, open-label, single ascending dose study. After being informed about the study and potential risks, all patients given written informed consent will undergo a screening to determine eligibility for study entry. Each subject will be enrolled in one of the three sequential cohorts, comprising one single dose of NEX-22A liraglutide injection. Each cohort will have a sentinel participant. NEX-22A will be administered in sequential cohorts. Before initiating a new dose cohort, safety, tolerability and PK data for all treated subjects must have been reviewed by the dose escalation committee. Blood samples for PK analysis will be withdrawn at specified timepoints over a period of 36 days

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent obtained before any trial-related activities. Trial-related activities are any procedures that would not have been done during normal management of the subject.
2. Male or female subject with type 2 diabetes mellitus.
3. Metformin therapy without change in dose for the last 3 months.
4. Age between 18 and 65 years, both inclusive.
5. Body Mass Index (BMI) between 18.5 and 35.0 kg/m^2, both inclusive.
6. HbA1c > 6.5% and <= 9.0%.
7. Diabetes duration of at least 1 year.

Exclusion Criteria:

1. Known or suspected hypersensitivity to the IMP or any of the excipients or to any component of the IMP formulation.
2. Previous participation in this trial. Participation is defined as being dosed.
3. Receipt of any medicinal product in clinical development within 30 days or at least 5 half-lives of the related substances and their metabolites (whichever is longer) before enrolment in this trial.
4. History of multiple and/or severe allergies to drugs or foods or a history of severe anaphylactic reaction.
5. Any history or presence of cancer except basal cell skin cancer or squamous cell skin cancer as judged by the investigator.
6. Clinically relevant comorbidity, capable of constituting a risk for the subject when participating in the trial or of interfering with the interpretation of data.
7. Signs of acute illness as judged by the investigator.
8. Any serious systemic infectious disease during four weeks prior to first dosing of the trial drug, as judged by the investigator.
9. Subjects with dermatological conditions, tattoos or large scars on the abdomen that would limit the evaluation of local tolerability, as judged by the investigator.
10. Clinically significant abnormal values for haematology, biochemistry, coagulation, or urinalysis at screening as judged by the investigator.
11. Systolic blood pressure < 90 mmHg or >160 mmHg and/or diastolic blood pressure < 50 mmHg or > 95 mmHg at screening (one repeat test will be acceptable in case of suspected white-coat hypertension).
12. Heart rate at rest (as measured in vital sign assessment at screening) outside the range of 50-90 beats per minute.
13. Clinically significant abnormal standard 12-lead electrocardiogram (ECG) after 5 minutes resting in supine position at screening, as judged by the investigator.
14. Proliferative retinopathy or maculopathy as judged by the investigator based on a recent (<1.5 years) ophthalmologic examination.
15. Severe neuropathy, in particular autonomic neuropathy, as judged by the investigator.
16. Former or current use of liraglutide or any other GLP-1 receptor agonists (exenatide, semaglutide) except for the use in clinical trials.
17. Current use of any insulin or sulfonylureas.
18. Significant history of alcoholism or drug abuse as judged by the investigator or consuming more than 24.0 grams alcohol/day (for males), 12.0 grams alcohol/day (for females) on average.
19. A positive result in the alcohol and/or urine drug screen at the screening visit.
20. Smoking more than 5 cigarettes or the equivalent per day.
21. Inability or unwillingness to refrain from smoking and use of nicotine substitute products one day before and during the inpatient period.
22. Tested positive for hepatitis Bs antigen.
23. Tested positive for hepatitis C antibodies. (Presence of hepatitis C antibodies will not lead to exclusion if liver function tests are normal and a hepatitis C polymerase chain reaction is negative).
24. Positive result to the test for HIV-1/2 antibodies or HIV-1 antigen.
25. Any medication (prescription and non-prescription drugs) within 14 days before IMP administration and/or anticoagulant therapy.
26. Blood donation or blood loss of more than 500 mL within the last 3 months.
27. Mental incapacity, unwillingness or language barriers precluding adequate understanding or co-operation.
28. Committed to an institution by virtue of an order issued either by the judicial or the administrative authorities.
29. Women of childbearing potential.
30. Trial site personnel directly affiliated with this trial and their immediate families (spouse, biological or legal guardian, child, or sibling).
31. The investigator considers a subject as unsuitable for inclusion in the trial for any other reason.

Explanatory note on Exclusion Criterion 25: Exceptions are stable doses of metformin, SGLT2-blockers, low dose aspirin, antihypertensives, statins, thyroid hormones or occasional use of paracetamol or ibuprofen, and ,if female, with the exception of menopausal hormone replacement therapy.

Explanatory note on Exclusion Criterion 29: A woman is considered of childbearing potential following menarche and until becoming postmenopausal unless permanently sterile due to hysterectomy, or bilateral salpingectomy, or bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-05-27 (Actual); Primary Completion 2025-07-18 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
To evaluate the PK profile of liraglutide after single ascending doses of NEX-22A in subjects with stable type 2 diabetes | From administration of study drug until 36 days
  Blood samples will be collected in order to calculate a PK profile. Maximum observed plasma concentration (Cmax)
To evaluate the PK profile of liraglutide after single ascending doses of NEX-22A in subjects with stable type 2 diabetes | From administration of study drug until 36 days
  Blood samples will be collected in order to calculate a PK profile. Time of occurrence of Cmax (Tmax)
To evaluate the PK profile of liraglutide after single ascending doses of NEX-22A in subjects with stable type 2 diabetes | From administration of study drug until 36 days
  Blood samples will be collected in order to calculate a PK profile. occurrence of Area under the plasma concentration vs. time curve (AUC) from time 0 to 8 hours (AUC0-8h)
To evaluate the PK profile of liraglutide after single ascending doses of NEX-22A in subjects with stable type 2 diabetes | From administration of study drug until 36 days
  Blood samples will be collected in order to calculate a PK profile. AUC from time 0 to 12 hours (AUC0-12h)
To evaluate the PK profile of liraglutide after single ascending doses of NEX-22A in subjects with stable type 2 diabetes | From administration of study drug until 36 days
  Blood samples will be collected in order to calculate a PK profile. AUC from time 0 to 24 hours (AUC0-24h)
To evaluate the PK profile of liraglutide after single ascending doses of NEX-22A in subjects with stable type 2 diabetes | From administration of study drug until 36 days
  Blood samples will be collected in order to calculate a PK profile. AUC from time 0 to 72 hours (AUC0-72h)
To evaluate the PK profile of liraglutide after single ascending doses of NEX-22A in subjects with stable type 2 diabetes | From administration of study drug until 36 days
  Blood samples will be collected in order to calculate a PK profile. AUC from time 0 to 7 days (AUC0-7days)
To evaluate the PK profile of liraglutide after single ascending doses of NEX-22A in subjects with stable type 2 diabetes | From administration of study drug until 36 days
  Blood samples will be collected in order to calculate a PK profile. AUC from 0 to time of last measurable plasma concentration (AUClast)
To evaluate the PK profile of liraglutide after single ascending doses of NEX-22A in subjects with stable type 2 diabetes | From administration of study drug until 36 days
  Blood samples will be collected in order to calculate a PK profile. AUC from time 0 to infinity (AUCinf)
To evaluate the PK profile of liraglutide after single ascending doses of NEX-22A in subjects with stable type 2 diabetes | From administration of study drug until 36 days
  Blood samples will be collected in order to calculate a PK profile. Terminal elimination half-life (T1/2)

SECONDARY OUTCOMES:
Number of subjects with treatment-related adverse events a assessed by frequency | From administration of study drug until 36 days
  Number of events.Descriptive individual data.
Number of subjects with treatment-related adverse events a assessed by seriouness | From administration of study drug until 36 days
  Seriousness of adverse events. Descriptive individual data.
Number of subjects with treatment-related adverse events a assessed by intensity | From administration of study drug until 36 days
  Intensity of adverse events. Descriptive individual data.
Number of subjects with treatment-related adverse events a assessed by relationship to study treatment | From administration of study drug until 36 days
  Relationship to study treatment. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the systolic blood pressure at 36 days | From administration of study drug until 36 days
  Measured in mmHg after 10 minutes supine rest. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in in the diastolic blood pressure at 36 days | From administration of study drug until 36 days
  Measured in mmHg after 10 minutes supine rest. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the ECG parameter PQ/PR at 36 days | From administration of study drug until 36 days
  Measured in ms in supine position after 5 minutes of rest using an ECG machine. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the ECG parameter QRS at 36 days | From administration of study drug until 36 days
  Measured in ms in supine position after 5 minutes of rest using an ECG machine. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the ECG parameter QT at 36 days | From administration of study drug until 36 days
  Measured in ms in supine position after 5 minutes of rest using an ECG machine. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the ECG parameter QTcB at 36 days | From administration of study drug until 36 days
  Measured in ms in supine position after 5 minutes of rest using an ECG machine. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the ECG parameter heart rate at 36 days | From administration of study drug until 36 days
  Measured in ms in supine position after 5 minutes of rest using an ECG machine. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the haematology blood parameters measurements at 36 days | From administration of study drug until 36 days
  Blood samples for the analysis of haematology parameters will be collected through venepuncture or an indwelling venous catheter. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the clinical chemistry blood laboratory measurements at 36 days | From administration of study drug until 36 days
  Blood samples for the analysis of clinical chemistry parameters will be collected through venepuncture or an indwelling venous catheter. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the coagulation blood laboratory measurements at 36 days | From administration of study drug until 36 days
  Blood samples for the analysis of coagulation parameters will be collected through venepuncture or an indwelling venous catheter. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in plasma glucose measurement at 36 days | From administration of study drug until 36 days
  Blood samples for the analysis of plasma glucos will be collected through venepuncture or an indwelling venous catheter. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the physical examination of the head at 36 days | From administration of study drug until 36 days
  Physical examination including assessment of the head. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the physical examination of the eyes at 36 days | From administration of study drug until 36 days
  Physical examination including assessment of the eyes. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the physical examination of the ears at 36 days | From administration of study drug until 36 days
  Physical examination including assessment of the ears. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the physical examination of the nose at 36 days | From administration of study drug until 36 days
  Physical examination including assessment of the nose. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the physical examination of the throat at 36 days | From administration of study drug until 36 days
  Physical examination including assessment of the throat. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the physical examination of the skin and mucosae at 36 days | From administration of study drug until 36 days
  Physical examination including assessment of the skin and mucosae. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the physical examination of the tyroid at 36 days | From administration of study drug until 36 days
  Physical examination including assessment of the tyroid. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the physical examination of the neurological status at 36 days | From administration of study drug until 36 days
  Physical examination including assessment of the neurological status. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the physical examination of the lungs at 36 days | From administration of study drug until 36 days
  Physical examination including assessment of the lungs. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the physical examination of the cardiovascular system at 36 days | From administration of study drug until 36 days
  Physical examination including assessment of the cardiovascular system including inspection, palpation, and auscultation.Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the physical examination of the gastrointestinal system incl mouth at 36 days | From administration of study drug until 36 days
  Physical examination including palpation of the gastrointestinal system incl mouth check. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the physical examination of the lymfh nodes incl mouth at 36 days | From administration of study drug until 36 days
  Physical examination including palpation of the lymfh nodes. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the musculoskeletal system at 36 days. | From administration of study drug until 36 days
  Physical examination of the musculoskeletal system. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in local tolerability i.e skin reactions assessed by visual inspection. | From administration of study drug until 36 days
  Visual inspection. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in local tolerability i.e skin reactions assessed by photography. | From administration of study drug until 36 days
  Photography of injection site Descriptive individual data.

CONTACTS AND LOCATIONS:
Overall Officials: Grit Andersen, MD, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH Hellersbergstr. 9 D-41460 Neuss
Locations (1):
- Profil, Neuss, Germany

IPD SHARING:
Plan to Share IPD: No